CLINICAL TRIAL: NCT02880501
Title: Safety and Effectiveness of Proximal Femoral Nail Antirotation for the Treatment of Intertrochanteric Femoral Fracture: Study Protocol for a Prospective Case Series
Brief Title: Safety and Effectiveness of Proximal Femoral Nail Antirotation for the Treatment of Intertrochanteric Femoral Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chaohu Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Junjie Xu, Associate Chief Physician, Chaohu Hospital of Anhui Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChaohuH_001
Record Dates: First submitted 2016-08-18; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Intertrochanteric Femoral Fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- proximal femoral nail antirotation (Experimental): Twenty patients with intertrochanteric femoral fracture scheduled will undergo proximal femoral nail antirotation (PFNA) implantation.
  Interventions: Device: proximal femoral nail antirotation

INTERVENTIONS:
Device: proximal femoral nail antirotation — Twenty patients with intertrochanteric femoral fracture scheduled to undergo proximal femoral nail antirotation (PFNA) implantation.

SUMMARY:
Minimally invasive PFNA fixation for the treatment of intertrochanteric femoral fracture will be used in 20 patients within 2 years to objectively validate the safety and effectiveness of PFNA in the treatment of fracture of long tube-like bone.

DETAILED DESCRIPTION:
History and current status of related studies Intertrochanteric femoral fracture frequently occurs in the elderly that is often complicated by different levels of osteoporosis, and mostly belongs to unstable fractures. This disorder is also frequently complicated by various chronic diseases, which make patients have poorer surgical tolerance. Surgical treatment is the widely accepted treatment method of intertrochanteric femoral fracture because it can accelerate the recovery and reduce the complications caused by long-term bed time. Intertrochanteric femoral fracture is unstable and occurs mostly in the elderly, so surgical treatment should meet the requirements including less risk of wound infection, less intraoperative blood loss, great holding potential and strong stability of the implants, which contribute to early hip joint function exercise and facilitate recovery after surgery.

According to the design principle of orthopedic implants, intramedullary and extramedullary fixations are commonly used. Compared to extramedullary fixation, intramedullary fixation places fixators closer to the affected region, produces shorter moment arm of force, better shares the compression forces on the medial cortex of the femoral neck, exhibits higher shear resistance, and provides greater stabilization for complex fractures in the elderly.

Compared to Garmma nail, an AO (Association for Osteosynthesis) proximal femoral nail has an antirotation screw in the proximal end which ensures an elastic fixation of the fracture and reduces the complications such as femoral shaft fractures. Nevertheless, 2 screws should be installed in the femoral neck, which restricts the slippage between the main screw and the compression screw, thus partial loading will be delivered through antirotation screws, leading to occurrence of complications such as antirotation screw cutting and compression screw withdrawal.

Conventional internal fixation methods including implantations of dynamic hip screws, Gamma nails, and proximal femoral intramedullary nail exhibit unfavorable effects in the treatment of intertrochanteric femoral fracture, in particular those complicated by severe osteoporosis because these methods cannot achieve firm and reliable fixation with occasional nail head cutting and nail withdrawal. Therefore, AO/ASIF (Association for Osteosynthesis/Association for the Study of Internal Fixation) designed a novel antirotation intramedullary nail, which better reduces the abovementioned complications.

Proximal femoral nail antirotation (PFNA) is a device designed based on proximal femoral intramedullary nail and other intramedullary nails. This device is equipped with a spiral wide blade which exhibits obvious antirotation and angular shear stress abilities, greatly reducing complications and decreasing the possibility of surgical delay. Compared to conventional screw systems, PFNA provides stronger antirotation and anti-inversion abilities. For tapping of a spiral blade in the femoral neck, only lateral femoral cortex should be opened without a need to remove bone matrix. The spiral blade tapped in the femoral neck will produce compression to the bone in the femoral neck. Even though for patients with severe osteoporosis, the spiral blade in the femoral neck can produce firm anchoring force with the femoral neck. Compared with screw fixation, a spiral blade exhibits a larger rotational torque, requires a smaller strength to be pulled out, and does not need additional screws tapped in the femoral neck, so the latter is easier to be operated. The PFNA has a medial-lateral angle of 6°, this allows insertion at the tip of the greater trochanter. The distal diameter of the PFNA is relatively small, and its eccentricity is reduced compared to that of intramedullary nails, which is more suitable to the anatomical morphology of proximal femoral medullary cavity. The locking pores of the PFNA at its distal tip include round static and oval-shaped dynamic types. Vertical installation of screws is considered dynamic interlocking and oblique installation of screws static interlocking. From the perspective of design, PFNA exhibits better biomechanical stability and shows advantages in duration of surgery, intraoperative blood loss, failure rate of surgery and overall complications over than internal fixation methods.

PFNA for the treatment of intertrochanteric femoral fracture in many cases has been reported, but related studies are mainly retrospective case series, and a few retrospective randomized controlled trials are reported.

Features different from other related studies Progress: PFNA is a device designed based on modification of Garmma nail and it integrates the advantages of a dynamic hip screw (DHS) used for extramedullary fixation and an intramedullary fixation device. PFNA exhibits more advantages over DHS, including (1) smaller stress shielding, being more conducive to fracture healing, and reduced cut-out phenomenon; (2) better shares the compressive stress of medial femur, leading to lower incidence of hip deformity. Both proximal femoral intramedullary nail and PFNA belong to intramedullary nails, but the latter exhibits the following advantages: (1) one assembly can achieve antirotation and angular stability; (2) the wide blade at the tip can compress as much peripheral matrix as possible, in particular under the circumstance of osteoporosis, exhibiting better holding potential; (3) the blade of PFNA is more closely attached to the matrix, which strengthens the stabilization of implant and prevents against rotation and varus deformity; (4) biomechanical tests have confirmed that the spiral blade can greatly increase shearing capacity; (5) spiral blades are implanted via a lateral incision and internal fixation has the features including minimal wound, less bleeding, satisfied reduction, rapid recovery, highly stable fractured stumps, being more conducive to early exercise, avoidance of prolonged force arm caused by extramedullary fixation, increased shear stress in the proximal femur, which greatly reduce the possibility of failure of internal fixation.

Feasibility: Intramedullary nail for the treatment of long bone fracture has been widely used in the clinic and expert consensus has been achieved. The novel PFNA for the treatment of interchochanteric femoral fracture in the elderly produces minimal wound, is easily performed, and is therefore highly feasible in the clinic. Our team has been ready for performing this project from various perspectives: (1) Personnel: This project will be equipped with 2 chief physicians, 2 associate chief physicians, 3 attending physicians, 2 resident physicians, and 1 graduate student. Our team has a strong clinical and scientific research capacity. (2) Techniques: our team has performed open or closed reduction and intramedullary nail fixation in many patients, so we are experienced, can provide sophisticated surgical skills in orthopedic trauma and joint surgery. (3) Equipment: The study setting has been equipped with orthopedic traction bed, X-ray, CT, MR scanners and other large equipments. All of these can provide hardware and software support.

Safety: Under fluoroscopic guidance, closed reduction will be followed by minimally invasive intramedullary nail fixation, which can effectively avoid vessel and nerve injury.

Data collection, management, analysis and open access Data collection: According to trial design type and requirement, a table will be developed to record trial data. The recorded data will be input into an electronic database using a double-data entry strategy by trained professional staff.

Data management: Information accuracy will be checked when all recruited patients are followed up. The database will be locked by the research in charge and will not be altered. All information relating to this trial will be preserved by Chaohu Hospital of Anhui Medical University, China.

Data analysis: The electronic database will be fully disclosed to a professional statistician for statistical analysis.

Data open access: Anonymized trial data will be published at www.figshare.com.

Statistical analysis Statistical analysis will be performed using SPSS19.0 software. The normally distributed continuous variables will be expressed as the mean ± standard deviation, and those non-normally distributed variables will be expressed as median and quartile. The categorical variables will be expressed as counts and the percentage. Paired t test or Wilcoxon test (paired samples) will be used for comparison of continuous variables between prior to and after PFNA implantation and the chi-square test for comparison of categorical variables between prior to and after PFNA implantation. A level of P < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Intertrochanteric femoral fracture diagnosed by anterior-posterior and lateral X-ray images, CT and MRI scans
* Types II-IV intertrochanteric femoral fracture in Evans-Jensen classification (Fung et al., 2007)
* Osteoporosis-caused intertrochanteric femoral fracture
* Fresh closed fracture (surgery performed within 2 weeks after fracture)
* Surgery performed for the first time after fracture
* Healthy and able to tolerance to anesthesia and surgery
* Age >18 years
* Provision of informed consent about participation and trial procedure

Exclusion Criteria:

* Not suitable to undergo internal fixation (such as severe osteoarthritis, rheumatoid arthritis and pathological fracture)
* Has installed other auxiliary devices in injured hip joint
* Infection of tissue around the hip joint
* With bone metabolism disorders besides osteoporosis, such as renal osteodystrophy and osteomalacia
* With heart, lung, brain and other systemic diseases
* With advanced malignant tumor
* Recently suffering from cerebral hemorrhage, myocardial infarction, and failure of important organs which are difficult to be corrected
* With injured limb deep venous thrombosis
* With mental disorders
* Unable to tolerance to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Complications | 6 months after surgery
  pains on the affected region, wound nonunion, incision infection

SECONDARY OUTCOMES:
Fracture healing | baseline, at 3 and 6 months after surgery
  evaluated by X-ray images
Hip joint function | baseline, at 3 and 6 months after surgery
  evaluated by Harris hip scores
Patient's quality of life | baseline, at 3 and 6 months after surgery
  evaluated by EuroQol five dimensions questionnaire (EQ-5D)
Barthel Index of Activities of Daily Living (Barthel ADL Index) | baseline, at 3 and 6 months after surgery
  Barthel ADL Index is used to evaluate patient's activities of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Junjie Xu, MD, Principal Investigator — Chaohu Hospital of Anhui Medical University

IPD SHARING:
Plan to Share IPD: Undecided